CLINICAL TRIAL: NCT06413030
Title: Slow Gait Speed as an Indicator of Overweight, Dynapenic Obesity and Sarcopenic Obesity in Elderly People in the Community
Acronym: SGSF
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Americas (Other)
Responsible Party: Principal Investigator, Karen Córdova-León, Academic Leader, University of Americas
Other Study IDs: CEC_FP_2023023
Record Dates: First submitted 2024-05-06; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Frailty; Obesity; Sarcopenia; Sarcopenic Obesity; Gait Speed
Keywords: aged; Aged, 80 and over
MeSH Terms: conditions — Frailty; Obesity; Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community-dwelling older adults: Persons over 60 years of age attending primary health care centers in the Bio Bio Region of Chile.
  Interventions: Diagnostic Test: 10 Meter Walk Test

INTERVENTIONS:
Diagnostic Test: 10 Meter Walk Test — Gait Speed Test

SUMMARY:
The goal of this observational study is to evaluate the relationship of gait speed with dynapenic or sarcopenic obesity in community-dwelling older people. The main questions it aims to answer are:

* Is slow walking speed related to overweight in older people in the community?
* Is slow walking speed related to dynapenic obesity in older people in the community?
* Is gait speed related to sarcopenic obesity in older people in the community?

Participants will answer a clinical interview to obtain sociodemographic data and will perform the following clinical tests: (1) 10-meter walk test, (2) Anthropometric measurement; (3) Handgrip dynamometry test, (4) Standing dynamometry test and (5) Physical functionality questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 60 years of age
* Female and male
* Self-sufficient in the instrumental activities of daily living
* Subjects with or without drug consumption, capable of carrying out the activity of walking independently or dependent on technical aids.

Exclusion Criteria:

* Subjects with acute musculoskeletal injuries of the lower extremity.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Older people who live in the community and attend primary health care centers in the Bio Bio Region of Chile.
Sampling Method: Non-Probability Sample
Enrollment: 383 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Gait Speed | Month 1
  A well-lit, unobstructed flat corridor with an extension of 10 meters is used for the test. Ground markings are added at 0 and 10 meters apart, with 2 meters start (acceleration) and 2 meters end (deceleration) added to allow participants room to accelerate and decelerate their walk outside the data collection area to help reduce the gait variability introduced during these phases. Subjects were instructed to walk at a usual and comfortable speed, without running or stopping. Subjects are allowed to use usual technical aids for walking, including walkers or canes if required. Chronometers based on smartphones to time the route between the second and third line of the route that consists of the 10 timed meters. The stopwatch records the time at which the subject's toe crossed the line. This sequence is repeated three times with 1 minute rest periods. The average of the three trials is used to determine the walking speed.
Anthropometric measures | Month 1
  Biospace Inbody: Individuals are placed in a standing position with 30º flexion of the scapulo-humeral joint. 8 electrodes are used located on: feet (metatarso-calcaneus) and hands (metacarpals 2nd-5th finger and phalanx of the thumb). The induction frequency is assessed with 6 different intensities (1, 5, 50, 250, 500 kHz and 1 MHz), with a fat mass estimation sensitivity of 0.1 kg (0.1%). From this measurement we obtain: percentage of muscle mass, percentage of general fat, percentage of visceral fat and bone weight.
Handgrip dynamometry | Month 1
  To evaluate manual muscle strength, the Baseline handgrip dynamometer will be used. The assessment is carried out with the subject in a seated position in a chair without armrests, with the back and feet adequately supported on the floor while the hips and knees are at 90°. The position was with shoulders adducted and neutrally rotated, elbows flexed at 90° and forearms in a neutral position. We began by evaluating the dominant hand by positioning the wrist between 15 and 30° of extension and between 0° and 15° of ulnar deviation. The dynamometer must be used in a vertical position, and parallel to the forearm, while the participant grips the handle with a thumbs up. 3 repetitions were performed for each limb, obtaining an average of the measurements, the grip time will be 3 to 6 seconds with a rest time of 1 minute, using the best value for data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Córdova-León, PT, Principal Investigator — Academic
Locations (1):
- Universidad de las Américas, Concepción, Chile

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR
URL: https://drive.google.com/drive/folders/1MfnO_AQUoTkjYsOZ1DKZ8vQrZhxsQiyN?usp=sharing